CLINICAL TRIAL: NCT04063124
Title: Pilot Study to Investigate the Safety and Feasibility of Senolytic Therapy to Modulate Progression of Alzheimer's Disease (SToMP-AD)
Brief Title: Senolytic Therapy to Modulate Progression of Alzheimer's Disease
Acronym: SToMP-AD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mitzi Gonzales, PhD, Associate Professor, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC20190222H
Record Dates: First submitted 2019-08-01; First posted 2019-08-21 (Actual); Results first posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Alzheimer Disease
Keywords: Dementia; Alzheimer; Cognitive decline; dasatinib
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction | interventions — Dasatinib; Quercetin

STUDY DESIGN:
Intervention Model Description: This study is an open-label pilot study of intermittent D+Q to measure its target engagement in CSF and blood, and to establish the feasibility and safety of D+Q treatment in older adults with early stage AD as initial proof-of-concept for a larger Phase 2 clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intermittent D+Q (Experimental): Senolytic treatment in 5 individuals with early AD to determine levels of drug that reach the central nervous system (CNS) by collecting cerebral spinal fluid (CSF), and begin collecting initial data on target engagement of senescent cells, AD-related markers, and AD-relevant outcomes for future trials.
  Interventions: Drug: Dasatinib + Quercetin

INTERVENTIONS:
Drug: Dasatinib + Quercetin — Intermittent D+Q administered for 2 days on/14 days off for 12 weeks (6 cycles)
  Other Names: D+Q

SUMMARY:
The purpose of this pilot study is to evaluate whether a combination of two drugs, dasatinib (D) and quercetin (Q) [D+Q], penetrate the brain using cerebrospinal fluid (CSF) in older adults with early Alzheimer's disease (AD). This combination of drug therapy has been shown to affect dying cells in humans with other chronic illnesses and in Alzheimer's mice models. The study team want to know if this combination of medications will reach the brain in order to evaluate if this intervention may be effective for treating AD symptoms in future studies. This is also known as a "proof of concept" study.

DETAILED DESCRIPTION:
Up to 40 potential candidates will be pre-screened to identify eligible men and women ages 65 years and over with a clinical diagnosis of early AD on a stable dose of cholinesterase inhibitors for at least 3 months (for example, Aricept).

Eligible participants will undergo laboratory assessments of blood and urine, receive study medications over a twelve week period, and complete pre- and post-treatment testing including: an MRI for digital imaging of the brain; lumbar puncture to obtain cerebrospinal fluid; memory and thinking assessments; quality of life questionnaires; and tests of walking, balance and strength, all of which will be done for research purposes only.

Participants must be accompanied by a Legally Authorized Representative and have no travel plans for 4-5 months that would interfere with study visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 years or above.
2. Clinical diagnosis of AD (MoCA 10-20 and Clinical Dementia Rating Scale/CDR = 1) on a stable dose of cholinesterase inhibitors for at least three months
3. Body Mass Index (BMI) within range of 19 - 35 kg/ m2
4. Labs: Normal blood cell counts without clinically significant excursions (WBCs: 4,500-10,500 cells/mcL; absolute neutrophil count: 1,800-8,700 cells/mcL; platelets: 140-450 K/uL; hemoglobin 12.0-17.5 grams/dL); liver and renal function (AST 10-40 IU/L, total bilirubin 0.1-1.4 mg/dl); cholesterol (<240 mg/dl), triglycerides (<300 mg/dl), and glucose control (HbA1c < 7%). PT/PTT/INR within normal limits
5. Participants must be accompanied by a Legally Authorized Representative designated to sign informed consent and to provide study partner reported outcomes at all remaining visits
6. Participants must have no plans to travel over the next 4-5 months that interfere with study visits following consent

Exclusion Criteria:

1. Hearing, vision, or motor deficits despite corrective devices;
2. Alcohol or drug abuse;
3. MRI contraindications;
4. Myocardial infarction, angina, stroke or transient ischemic attack in the past 6 months; QT interval >440 on ECG will not be enrolled. Chronic heart failure will be exclusionary;
5. Participants with coagulation disorders;
6. Neurologic, musculoskeletal, or other condition that limits subject's ability to complete study physical assessments;
7. Uncontrolled diabetes (HbA1c > 7% or the current use of insulin);
8. Current or chronic history of liver disease, or known hepatic or biliary abnormalities;
9. Use of anti-arrhythmic medications known to cause QTc prolongation, anti-platelet or anti-coagulant medication;
10. Current use of quinolone antibiotics.
11. Poorly controlled blood pressure (systolic BP>160, diastolic BP>90 mmHg).
12. Active inflammatory, autoimmune, infectious, hepatic, gastrointestinal, malignant, and psychiatric disease.
13. History of or MRI-positive for any space occupying lesion, including mass effect or abnormal intracranial pressure, which would indicate contraindication to lumbar puncture

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-02-14 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Musi, MD, Principal Investigator — UT Health San Antonio
Locations (1):
- Glenn Biggs Institute for Alzheimer's & Neurodegenerative Diseases, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: At study completion
Access Criteria: Through journal publication

REFERENCES:
- [Derived] Garbarino VR, Palavicini JP, Melendez J, Barthelemy NR, He Y, Kautz TF, Lopez-Cruzan M, Mathews JJ, Xu P, Zhang B, Saliba A, Ragi N, Sharma K, Mason D, Johnson S, Hendrix S, Craft S, Petersen RC, Espindola-Netto JM, Xue A, Tchkonia T, Kirkland JL, Salardini A, Musi N, Bateman RJ, Gonzales MM, Orr ME. Evaluation of exploratory fluid biomarkers from a phase 1 senolytic trial in mild Alzheimer's disease. Neurotherapeutics. 2025 Jul;22(4):e00591. doi: 10.1016/j.neurot.2025.e00591. Epub 2025 Apr 23. PMID 40274471
- [Derived] Andrews TD, Day GS, Irani SR, Kanekiyo T, Hickson LJ. Uremic Toxins, CKD, and Cognitive Dysfunction. J Am Soc Nephrol. 2025 Jun 1;36(6):1208-1226. doi: 10.1681/ASN.0000000675. Epub 2025 Feb 26. PMID 40009460
- [Derived] Garbarino VR, Palavicini JP, Melendez J, Barthelemy N, He Y, Kautz TF, Lopez-Cruzan M, Mathews JJ, Xu P, Zhan B, Saliba A, Ragi N, Sharma K, Craft S, Petersen RC, Espindola-Netto JM, Xue A, Tchkonia T, Kirkland JL, Seshadri S, Salardini A, Musi N, Bateman RJ, Gonzales MM, Orr ME. Evaluation of Exploratory Fluid Biomarker Results from a Phase 1 Senolytic Trial in Mild Alzheimer's Disease. Res Sq [Preprint]. 2024 Mar 8:rs.3.rs-3994894. doi: 10.21203/rs.3.rs-3994894/v1. PMID 38496619
- [Derived] Gonzales MM, Garbarino VR, Kautz TF, Palavicini JP, Lopez-Cruzan M, Dehkordi SK, Mathews JJ, Zare H, Xu P, Zhang B, Franklin C, Habes M, Craft S, Petersen RC, Tchkonia T, Kirkland JL, Salardini A, Seshadri S, Musi N, Orr ME. Senolytic therapy in mild Alzheimer's disease: a phase 1 feasibility trial. Nat Med. 2023 Oct;29(10):2481-2488. doi: 10.1038/s41591-023-02543-w. Epub 2023 Sep 7. PMID 37679434
- [Derived] Sarkar P, Kumar A, Behera PS, Thirumurugan K. Phytotherapeutic targeting of the mitochondria in neurodegenerative disorders. Adv Protein Chem Struct Biol. 2023;136:415-455. doi: 10.1016/bs.apcsb.2023.02.013. Epub 2023 Mar 24. PMID 37437986
- [Derived] Gonzales MM, Garbarino VR, Marques Zilli E, Petersen RC, Kirkland JL, Tchkonia T, Musi N, Seshadri S, Craft S, Orr ME. Senolytic Therapy to Modulate the Progression of Alzheimer's Disease (SToMP-AD): A Pilot Clinical Trial. J Prev Alzheimers Dis. 2022;9(1):22-29. doi: 10.14283/jpad.2021.62. PMID 35098970
- [Derived] Gonzales MM, Krishnamurthy S, Garbarino V, Daeihagh AS, Gillispie GJ, Deep G, Craft S, Orr ME. A geroscience motivated approach to treat Alzheimer's disease: Senolytics move to clinical trials. Mech Ageing Dev. 2021 Dec;200:111589. doi: 10.1016/j.mad.2021.111589. Epub 2021 Oct 21. PMID 34687726

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects that were consented and passed screening
Period: Overall Study
Arm/Group | Intermittent D+Q
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Five participants enrolled in the intervention
Arm/Group | Intermittent D+Q
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 76 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Educational level [Count of Participants; unit: Participants]
  High school graduate | 2
  Some college | 1
  College degree or higher | 2

OUTCOME MEASURES:

1. Primary Outcome: Brain Penetrance of Dasatinib (D)
Description: Cerebrospinal Fluid (CSF) collected by lumbar puncture before and after 12 weeks of treatment to determine levels of drug that reach the central nervous system will be measured by high performance liquid chromatography/mass spectrometry (HPLC/MS)
Time Frame: Change from 0 to 12 weeks
Population: tandem mass spectrometry
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Intermittent D+Q
Number analyzed (Participants) | 5
ng/ml | 0.27 (0.19)

2. Primary Outcome: Brain Penetrance of Quercetin (Q)
Description: CSF collected by lumbar puncture before and after 12 weeks of treatment to determine levels of drug that reach the central nervous system using HPLC/MS
Time Frame: Change from 0 to 12 weeks
Population: tandem mass spectrometry
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Intermittent D+Q
Number analyzed (Participants) | 5
ng/ml | 0 (0)

3. Secondary Outcome: Alzheimer's Disease Marker - CSF Tau
Description: Cerebrospinal Fluid collected by lumbar puncture analyzed for level of tau proteins present in CSF
Time Frame: Change from 0 to 12 weeks
Population: total tau assessed by Simoa HD-X analyzer
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Intermittent D+Q
Number analyzed (Participants) | 5
pg/ml | -21 (35)

4. Secondary Outcome: Alzheimer's Disease Marker - CSF Amyloid Beta
Description: Cerebrospinal Fluid collected by lumbar puncture analyzed for level of amyloid beta proteins present in CSF
Time Frame: Change from 0 to 12 weeks
Population: Abeta 42 assessed using Simoa HD-X Analyzer
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Intermittent D+Q
Number analyzed (Participants) | 5
pg/ml | 78 (75)

5. Secondary Outcome: Senescence Marker IL-6 in CSF
Description: Laboratory measure of level of IL-6 found in CSF collected pre and post treatment
Time Frame: Change from 0 to 12 weeks
Population: Assessed using Meso-Scale Discovery platform
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Intermittent D+Q
Number analyzed (Participants) | 5
pg/ml | 0.37 (0.20)

6. Secondary Outcome: Senescence Marker P16 in CSF
Description: Laboratory measure of level of P16 found in CSF collected pre and post treatment
Time Frame: Change from 0 to 12 weeks
Population: Data were not collected for this outcome measure
Arm/Group | Intermittent D+Q
Number analyzed (Participants) | 0

7. Secondary Outcome: Electronic Gait Mapping Under Single and Dual-task Conditions
Description: Participants walk on a pressure-sensitive walkway to capture data on gait speed
Time Frame: Change from 0 to 12 weeks
Population: Data were not collected for this outcome measure
Arm/Group | Intermittent D+Q
Number analyzed (Participants) | 0

8. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: A test which scores the participant with score ranges between 0 and 30. A score of 26 or over is considered normal. Individuals with mild cognitive impairment score lower and individuals with Alzheimer's disease score even lower.
Time Frame: Change from 0 to 12 weeks
Population: Change in points out of 30
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Intermittent D+Q
Number analyzed (Participants) | 5
points | -0.20 (2.28)

ADVERSE EVENTS:
Time Frame: Baseline to 12 weeks
Arm/Group | Intermittent D+Q
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intermittent D+Q (N=5)
Fall (General disorders) | 1 (1) — Fall unrelated to intervention
Diarrhea (Gastrointestinal disorders) | 1 (1) — Mild diarrhea with same day resolution, unlikely to be related to intervention
Urinary tract infection (Renal and urinary disorders) | 2 (2) — Mild symptoms, unlikely to be related to intervention
Hypoglycemia (Endocrine disorders) | 1 (1) — Moderate, possibly related to intervention
Hematuria (Renal and urinary disorders) | 1 (1) — Prior to intervention administration, not related to intervention
Emesis (Gastrointestinal disorders) | 1 (1) — Mild with same day resolution, unlikely to be related to intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT04063124/Prot_SAP_000.pdf